CLINICAL TRIAL: NCT01388192
Title: Effects of Pancreaticoduodenectomy on Glucose Metabolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201104028RC
Record Dates: First submitted 2011-06-23; First posted 2011-07-06 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus; Glucose Intolerance
Keywords: Pancreaticoduodenectomy; diabetes; sugar metabolism
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Receiving pancreaticoduodenectomy

SUMMARY:
Pancreaticoduodenectomy (PD) involves removing the head of pancreas, duodenum, common bile duct, gall bladder, and/or distal stomach. In general, the postoperative changes are thought to be moderately severe, and about 20% of these patients go on to develop new clinical diabetes. PD-related factors of glucose metabolism will include removal of half of the pancreatic endocrine tissue, exclusion of the proximal small intestine, postoperative weight loss (on average, ~8% of body weight), and removal of putative diabetogenic factor in resected neoplasm. However, effect of removal of duodenum on glucose metabolism after PD has never been studied. The investigators plan to examine this issue by comparing fasting plasma levels of insulin, fasting plasma glucose, C-peptide, HbA1C, HOMA-insulin resistance, GLP-1 response after a standard meal, and body mass index (BMI) of patients before and after PD.

DETAILED DESCRIPTION:
Questionaire All studied patients will be requested to self-complete a detailed questionnaire that collects information on demographic data, including usual adult height and weight, and history of DM in first-degree relatives. Existing medical conditions, including DM, duration of these medical problems, and current medications will also be inquired. The database will also include details of weight measured at the time of recruitment and body mass index (BMI), calculated as weight (kg)/height2 (m2). All studied patients will have FBG levels measured. Patients receiving prescription antidiabetic medications for previously diagnosed DM will be classified as having DM regardless of their FBG value. Among patients not reporting treatment for DM, classification of DM status will be based on the American Diabetes Association criteria; patients will be classified as having DM if the FBG level is ≧126 mg/dL (7 mmol/L), as having impaired fasting glucose (IFG) if their FBG is between 100 and 125 mg/dL (5.6-6.9 mmol/L), and as having normal fasting glucose (NFG) if their FBG value is ≦99 mg/dL (5.5 mmol/L).

After withdrawal of anti-diabetic medications for 12 h, the patients were asked to fast overnight for 12 h, then were given 200 ml of formula (220kcal, 14g of protein, 28 g of carbohydrates, and 5 g of fat; Modifast, Stocksund, Sweden) within 10 min through a NG tube on post-operative day 5 (proximal feeding group [PFG]) and a jejunostomy feeding tube (distal feeding group [DFG]) on post-operative day 6. The below parameter will be checked, including

1. HOMA insulin resistance assessment (HOMA-IR)
2. GLP-1
3. GIP
4. C-peptide
5. Insulin
6. Glucose

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving pancreaticoduodenectomy

Exclusion Criteria:

* history of pancreatitis
* hepatic dysfunction (Child-Pugh > 2)
* renal dysfunction (serum creatinine concentration > 3 mg/L, hemodialysis, or both)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving pancreaticoduodenectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change of glucose metabolism after pancreaticoduodenectomy | on the post-operative day 5 and day 6
  Measurement of glucose, glucagon-like peptide-1, Measurement of insulin, C-peptide, and glucagon concentrations after meal test

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Wen Tien, M.D., Ph.D., Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan